CLINICAL TRIAL: NCT06591845
Title: A Single-Center, Randomized, Partially Double-Blind, Placebo- and Active-Controlled, Four-period Crossover, Thorough QT/QTc (TQT) Clinical Study to Evaluate the Effects of Ziresovir on Cardiac Repolarization in Healthy Subjects
Brief Title: Thorough QT/QTc (TQT) Clinical Study to Evaluate the Effects of Ziresovir on Cardiac Repolarization in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AK0529-3004
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: QT/QTc (TQT) Clinical Study
MeSH Terms: interventions — ziresovir; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: This clinical study will last for a total of 59 days, including a 26-day screening period, admission day (Day -2) preceding the first treatment period, 4 treatment periods with 8 days washout in-between and a safety follow-up period (7 ± 1 days after the last dose).
Who Masked: Participant
Masking Description: Partially Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment T (Therapeutic dose) (Experimental): The subjects will receive a ziresovir 125 mg as single dose on Day 1 (Period 1) or Day 9 (Period 2) or Day 17 (Period 3) or Day 25 (Period 4)
  Interventions: Drug: Ziresovir 125 mg
- Treatment ST (Supratherapeutic dose) (Experimental): The subjects will receive a ziresovir 500 mg as single dose on Day 1 (Period 1) or Day 9 (Period 2) or Day 17 (Period 3) or Day 25 (Period 4)
  Interventions: Drug: Ziresovir 500 mg
- Treatment P (Placebo) (Placebo Comparator): The subjects will receive a placebo as single dose on Day 1 (Period 1) or Day 9 (Period 2) or Day 17 (Period 3) or Day 25 (Period 4)
  Interventions: Drug: Placebo
- Treatment PC (positive control) (Active Comparator): The subjects will receive a moxifloxacin hydrochloride tablet 400 mg as single dose on Day 1 (Period 1) or Day 9 (Period 2) or Day 17 (Period 3) or Day 25 (Period 4)
  Interventions: Drug: Moxifloxacin hydrochloride tablet 400 mg

INTERVENTIONS:
Drug: Ziresovir 125 mg — Active Substance: Ziresovir, Pharmaceutical Form: Suspension, Route of Administration: Oral
  Arms: Treatment T (Therapeutic dose)
Drug: Ziresovir 500 mg — Active Substance: Ziresovir, Pharmaceutical Form: Suspension, Route of Administration: Oral
  Arms: Treatment ST (Supratherapeutic dose)
Drug: Placebo — Active Substance: Placebo, Pharmaceutical Form: Suspension, Route of Administration: Oral
  Arms: Treatment P (Placebo)
Drug: Moxifloxacin hydrochloride tablet 400 mg — Active Substance: Moxifloxacin hydrochloride Pharmaceutical Form: Tablet Route of Administration: Oral
  Arms: Treatment PC (positive control)

SUMMARY:
This is a single-center, randomized, partially double-blind, placebo and active-controlled, 4-period crossover design thorough QT/QTc (TQT) clinical study to evaluate the effects of ziresovir on cardiac repolarization in healthy subjects.

DETAILED DESCRIPTION:
This clinical study is a single-center, randomized, partially double-blind, placebo- and active-controlled, four-period crossover design, with healthy subjects comprising the enrolled population. Ziresovir and placebo will be administered in a double-blind manner, while moxifloxacin hydrochloride tablets will be administered in as open-label.

Thirty-two subjects meeting all inclusion criteria and none of the exclusion criteria will be randomized into 1 of 12 dosing sequences, each consisting of 4 periods with an 8-day washout period in-between.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily signed a written informed consent form.
2. Male or female; between 18 and 50 years old (inclusive).
3. Male subjects weighing ≥50 kg, female subjects weighing ≥45 kg, body mass index (BMI) between 19.0 and 30.0 kg/m2 (inclusive), BMI= weight (kg)/height2 (m2).
4. Healthy, as defined by no clinically significant or relevant abnormalities identified by vital signs, physical examination, laboratory examination items, ECG, and other trial-related examinations at screening, admission or baseline day of each period as assessed by the investigator.
5. The subject can communicate well with the investigator and is able to complete the study in compliance with the protocol.

Exclusion Criteria:

1. History of or evidence of clinically significant disorder, condition or disease not otherwise excluded that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
2. History of cardiovascular disease or risk factors for Torsade de Pointes (TdP) at screening, including but not limited to: unexplained syncope; heart failure; cardiomyopathy; hypertension; angina pectoris; myocardial infarction; hypokalemia; bradycardia or sick sinus syndrome; cardiac conduction abnormalities; personal or family history of long QT syndrome (LQTS); or family history of sudden death.
3. Known or suspected malignancy.
4. Known allergic reactions to study intervention (e.g., ziresovir or its drug excipients, moxifloxacin, fluoroquinolone antibiotics) or history of clinically significant multiple or severe drug allergies, food allergies.
5. Subjects who have donated blood or have had a blood loss ≥500 ml within 3 months prior to screening.
6. Subjects who have participated in a clinical trial evaluating an investigational drug or device within 30 days or 5 half-lives (whichever is longer) prior to screening.
7. History of substance abuse (e.g., alcohol, licit or illicit drugs) within 1 year prior to screening.
8. 12-lead ECG at screening or admission exceeding criteria: PR>220 ms, QRS>120 ms, HR< 50 bpm or >100 bpm, QTcF >450 ms (male and female) (The mean of 3 triplicate ECGs timepoint measurement); or ECG abnormalities that are considered by the investigator to be abnormal and clinically significant.
9. Systolic blood pressure (BP) > 140 mmHg or < 90 mmHg, or diastolic BP > 90 mmHg at screening or admission.
10. Serum potassium, calcium, or magnesium levels outside the normal range at screening or admission.
11. Positive blood alcohol test, positive urine cotinine test or positive urine drug abuse screening at screening or admission.
12. Engaged in strenuous exercise within 48 hours before randomization (e.g., marathon running, long-distance cycling, weightlifting).
13. Intake of caffeinated beverages or food within 48 hours before randomization or a history of high caffeine consumption (e.g., in the last 3 months drinking >5 cups of coffee/day).
14. History of alcoholism or regular alcohol consumption within 1 year prior to screening, defined as more than 14 units (male) or 7 units (female) of alcohol per week (1 unit =360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine).
15. Smoking or use of tobacco or nicotine-containing products within 6 months before screening.
16. Pregnant or lactating women or those with positive blood pregnancy test results.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline QTcF (ΔQTcF) | Before dosing (Baseline) through 48 hours after the dose on Day 1 in each treatment period
  The primary ECG endpoint is the change from baseline in the QT interval corrected for heart rate (HR) using the Fridericia method (ΔQTcF).

SECONDARY OUTCOMES:
Change from baseline in QTc | Before dosing (Baseline) through 48 hours after the dose on Day 1 in each treatment period
  Change from baseline in QTc using correction methods not chosen as the primary correction method if a substantial HR effect is observed
Change from baseline in HR, PR, and QRS | Before dosing (Baseline) through 48 hours after the dose on Day 1 in each treatment period
  Change-from-baseline in HR, PR and QRS (ΔHR, ΔPR and ΔQRS).
Incidence of treatment-emergent adverse events (TEAEs) and changes in laboratory safety tests, vital signs, and ECGs. | Up to Day 8 of each treatment period (up to 31 days)
  Incidence of treatment-emergent adverse events (TEAEs) and changes in laboratory safety tests, vital signs, and ECGs.
Treatment-emergent changes in ECG Morphology | Before dosing (Baseline) through 48 hours after the dose on Day 1 in each treatment period
  Treatment-emergent changes in ECG Morphology
Categorical outliers for QTcF/QTcI/QTcS, HR, PR, and QRS. | Before dosing (Baseline) through 48 hours after the dose on Day 1 in each treatment period
  Categorical outliers for QTcF/QTcI/QTcS, HR, PR, and QRS.
Maximum observed plasma concentration (Cmax) of ziresovir | Pre-dose within 1 hour and at 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, and 72 hours post-dose during each period
  PK parameters of ziresovir and its metabolites including maximum observed plasma concentration (Cmax).
Terminal elimination half-life (t1/2) of ziresovir. | Pre-dose within 1 hour and at 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, and 72 hours post-dose during each period.
  PK parameters of ziresovir and its metabolites including terminal elimination half-life (t1/2).
Area under the curve (AUC) of ziresovir. | Pre-dose within 1 hour and at 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, and 72 hours post-dose during each period.
  PK parameters of ziresovir and its metabolites including area under the curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: David Han, M.D., M.P.H, Principal Investigator — California Clinical Trials Medical Group

IPD SHARING:
Plan to Share IPD: No